CLINICAL TRIAL: NCT06453642
Title: Evaluation of a Simple-Prep Controlled Embolic (GPX Trial)
Brief Title: Evaluation of a Simple-Prep Controlled Embolic
Acronym: GPX
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fluidx Medical Technology, Inc. (Industry)
Collaborators: Bright Research Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLX-CL-5000
Record Dates: First submitted 2024-05-29; First posted 2024-06-11 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Embolization; Vascular Tumor; Renal Angiomyolipoma; Renal Cell Carcinoma; Bone Tumor; Portal Vein Embolization
Keywords: Embolization; Distal Embolization; Distal Vessel Penetration; Peripheral Vasculature
MeSH Terms: conditions — Vascular Neoplasms; Angiomyolipoma; Carcinoma, Renal Cell; Bone Neoplasms

STUDY DESIGN:
Intervention Model Description: The investigation is a single-arm, open-label, non-randomized, prospective, multicenter, multinational pivotal study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- GPX® Embolic Device (Experimental)
  Interventions: Device: GPX® Embolic Device

INTERVENTIONS:
Device: GPX® Embolic Device — Treatment includes distal embolization in the peripheral vasculature of vascular tumors, renal embolization, and portal vein branches

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of the GPX® Embolic Device when used as indicated for embolization requiring distal vessel penetration in 114 subjects in up to 25 investigational sites in the USA, New Zealand, and Canada.

DETAILED DESCRIPTION:
The investigation is a single-arm, open-label, non-randomized, prospective, multicenter, multinational pivotal study. Subjects will undergo distal embolization in the peripheral vasculature, including vascular tumors, renal embolizations, and portal vein branches, with the GPX® Embolic Device and will then be followed 30-days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years on the date of consent
2. Expected post-procedural lifespan of at least 30 days, in the opinion of the investigator, to allow for participation in all follow-up visits
3. Presents with need for peripheral embolization where there is a desire for distal vessel bed penetration including:

   * Vascular tumors (e.g., renal angiomyolipoma, renal cell carcinoma, bone tumors, bleeding tumors, and other vascular tumors)
   * Renal embolization
   * Portal vein branches
4. Informed consent granted by the patient or legally authorized representative
5. Willing and able to comply with the protocol-specified procedures and assessments

Exclusion Criteria:

1. Requires embolization for any of the following applications: a) Neurovasculature b) Coronary vasculature c) Hemorrhage due to trauma d) Non-tumoral focal/active bleeding sites (e.g., gastrointestinal tract, urinary tract, lung) e) Veins other than portal vein f) Aneurysms g) Endoleaks h) Vascular malformations i) Vessels for flow redistribution
2. Has undergone an embolization procedure within 30 days prior to consent
3. Presents with need for embolization where the risk of clinically significant infarction outweighs the benefit of distal penetration (e.g., gastrointestinal, uterine)
4. Embolization target is only intended for temporary occlusion (e.g., bioresorbable biologic embolic agents)
5. Known allergy or hypersensitivity to contrast media that cannot be adequately medicated
6. Pregnant, planning to become pregnant during the study period, or breastfeeding
7. Unresolved systemic infection or localized infection in the targeted region
8. Pre-operative laboratory tests and/or physical examination indicate abnormal results, which, in the opinion of the investigator, would clinically confound the study primary endpoints
9. Existing medical condition which, in the opinion of the investigator, may cause the subject to be intolerant of an occlusion procedure or non-compliant with the protocol or may confound the data interpretation
10. Subject is participating in another device, drug, or procedure clinical investigation and has not completed the study treatment or the other investigation clinically interferes with the endpoints of this study (post-approval registries are allowed as long as the investigator determines there is no clinical interference with study endpoints)
11. Vulnerable subject populations (e.g., incarcerated or cognitively challenged adults) 12. Patients with drug or alcohol dependency (within 6 months prior to study entry) that, in the opinion of the investigator, would interfere with safe delivery of the study treatment or with the interpretation of study results

Intra-procedural exclusion criteria:

13. Presence of persistent, flow-limiting vasospasm that is not responsive to chemical or mechanical interventions 14. Presence of collateral pathways potentially endangering normal territories during embolization 15. Blood flow precludes safe delivery of embolic material (e.g., arteriovenous shunting or high, unpredictable flow exists) 16. Anatomy that precludes advancement of the delivery device to target vessel embolization site or delivery of embolic material 17. Dissection in the target vessel 18. The delivery device has already been used with an ionic contrast agent (e.g., Conray® (iothalamate meglumine injection USP 60%), Guerbet)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Freedom from major adverse events (MAEs) | Index procedure through 30-day follow-up
  MAEs are defined as:
  * Nontarget embolization with ischemia in an unintended anatomical area
  * Systemic allergic and/or toxic reaction to the GPX Embolic Device
  * Catheter entrapment and/or breakage
  * Culture-proven abscess in target organ/tissue
  * Embolization-related death
Single binomial proportion of successful delivery of the GPX Embolic Device to the target vessel embolization site(s) | During procedure
  Determined by the investigator at the time of enrollment
Single binomial proportion of successful occlusion of flow immediately beyond the target vessel embolization site(s) | End of procedure
  Determined by the core lab via comparison of the pre- and final post-embolization images

SECONDARY OUTCOMES:
Occurrence of device-related adverse events (AE) through 30 days post-index procedure | 30-day follow-up
Occurrence of adjunctive embolization agent usage during the embolization procedure | End of procedure
Occurrence of catheter occlusion due to the GPX Embolic Material | End of procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Darcy, MD, Principal Investigator — Washington University School of Medicine
Locations (20):
- United States (15):
  - University of California San Diego Altman Clinical and Translation Research Institute, La Jolla, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Indiana University Hospital, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University - Barnes Jewish Hospital, St Louis, Missouri
  - Albany Medical Center, Albany, New York
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - University of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center - Interventional Radiology, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hosptial, Toronto, Ontario
  - Mount Sinai Hospital Toronto, Toronto, Ontario
- New Zealand (2):
  - Auckland City Hospital, Auckland
  - Christchurch Hospital, Christchurch

IPD SHARING:
Plan to Share IPD: No